CLINICAL TRIAL: NCT02997657
Title: Positive Psychotherapy for Smoking Cessation Enhanced With Text Messaging: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Truth Initiative (Other)
Responsible Party: Principal Investigator, Christopher W. Kahler, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01CA201262 (NIH)
Record Dates: First submitted 2016-12-05; First posted 2016-12-20 (Estimated); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychotherapy for Smoking Cessation (Experimental): Smoking cessation treatment that incorporates exercises and text messages derived from positive psychology interventions that are designed to boost positive moods, cognitions, and behaviors.
  Interventions: Behavioral: Positive Psychotherapy; Behavioral: Standard smoking cessation counseling
- Standard smoking cessation treatment (Active Comparator): Smoking cessation counseling that provides support and problem solving skills for avoiding smoking.
  Interventions: Behavioral: Standard smoking cessation counseling

INTERVENTIONS:
Behavioral: Positive Psychotherapy — Exercises designed to boost moods, positive behaviors, and positive cognitions.
  Arms: Positive Psychotherapy for Smoking Cessation
Behavioral: Standard smoking cessation counseling — Counseling designed to provide support and problem solving for smoking cessation

SUMMARY:
Positive Psychotherapy for Smoking Cessation (PPT-S) addresses an array of risk factors for poor smoking outcomes (low positive affect, depressive symptoms, and cynical cognitions), while also providing skills that may buffer against stress and negative affect. The overall objective of this project is to conduct a randomized controlled trial to test the efficacy of PPT-S, enhanced with text messaging, compared to a time-matched behavioral smoking cessation treatment. Participants in both treatment conditions will receive nicotine replacement therapy and a validated text-messaging intervention for smoking cessation that monitors progress in quitting smoking and extends smoking counseling outside of the individual face-to-face context.

ELIGIBILITY:
Inclusion Criteria:

1. be 18 years of age or older
2. smoke at least 5 cigarettes per day for longer than one year with no current regular use of other nicotine/tobacco products including e-cigarettes
3. have a baseline carbon monoxide level of at least 4 ppm
4. be willing to use the nicotine patch
5. report at least a 5 on a 0 to 10 scale rating the importance of quitting smoking (where 10 = extremely important);
6. have an active cell phone and be willing to send and receive text messages for the duration of the intervention.

Exclusion Criteria:

1. Contact study site for details

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kahler, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Partners Healthcare and Massachusetts General Hospital, Boston, Massachusetts
  - Center for Alcohol and Addiction Studies, Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment
Started | 140 | 131
Completed | 109 | 97
Not Completed | 31 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment | Total
Number analyzed (Participants) | 140 | 131 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (12.1) | 49.2 (12.0) | 49.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Self reported sex missing for one 1 participant
  Participants
    number analyzed (Participants) | 140 | 130 | 270
    Female | 78 | 71 | 149
    Male | 62 | 59 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 132 | 123 | 255
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 17 | 29
  White | 119 | 111 | 230
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 1 | 1 | 2
Fagerstrom test for cigarette dependence [Mean (Standard Deviation); unit: units on a scale] — Self report measure of cigarette dependence with scores ranging from 0 to 10, where 10 is the highest level of dependence.
  units on a scale | 5.1 (2.0) | 4.5 (2.1) | 4.8 (2.1)
CES-D Total Score [Mean (Standard Deviation); unit: units on a scale] — Center for Epidemiologic Studies-Depression Scale, total score. This 20-item scale has total scores ranging from 0-60 with higher scores indicating more severe depresssive symptoms. A score of 16 of greater is typically used to indicate possible major depressive disorder.
  units on a scale | 13.1 (10.0) | 12.1 (9.5) | 12.6 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Smoking Abstinence at 12 Weeks
Description: Self-reported smoking abstinence biochemically confirmed with CO and cotinine
Time Frame: 12 weeks
Population: 1 participant in the Positive Psychotherapy for Smoking Cessation condition died prior to the 12-week follow-up and was not included. All other participants were included in the primary analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment
Number analyzed (Participants) | 139 | 131
Participants | 29 | 25
Statistical Analysis 1: Comparison: Positive Psychotherapy for Smoking Cessation vs Standard Smoking Cessation Treatment; Test type: Superiority; p = 0.71, Chi-squared

2. Primary Outcome: 7-day Point Prevalence Smoking Abstinence at 26 Weeks
Description: Self-reported smoking abstinence biochemically confirmed with CO and cotinine
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment
Number analyzed (Participants) | 139 | 131
Participants | 27 | 27
Statistical Analysis 1: Comparison: Positive Psychotherapy for Smoking Cessation vs Standard Smoking Cessation Treatment; Test type: Superiority; p = 0.81, Chi-squared

3. Primary Outcome: 7-day Point Prevalence Smoking Abstinence at 52 Weeks
Description: Self-reported smoking abstinence biochemically confirmed with CO and cotinine
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment
Number analyzed (Participants) | 139 | 131
Participants | 27 | 28
Statistical Analysis 1: Comparison: Positive Psychotherapy for Smoking Cessation vs Standard Smoking Cessation Treatment; Test type: Superiority; p = 0.69, Chi-squared

4. Primary Outcome: Continuous Smoking Abstinence
Description: Self-reported continuous abstinence from cigarette smoking from quit date through the 52-week follow-up biochemically confirmed at 12, 26, and 52 weeks
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment
Number analyzed (Participants) | 139 | 131
Participants | 13 | 12
Statistical Analysis 1: Comparison: Positive Psychotherapy for Smoking Cessation vs Standard Smoking Cessation Treatment; Test type: Superiority; p = 0.96, Chi-squared

5. Secondary Outcome: Engagement in PPT-consistent Quitting Strategies
Description: Engaging in strategies consistent with the positive psychology exercises taught in the trial. Nine strategies are assessed on 1 to 5 scale with 5 reflecting greater use of the strategies. The total score is the average across the 9 item.
Time Frame: During treatment - weeks 1-4 after quit date
Population: Participants were asked these questions at the final session of counseling. Therefore only participants attending that session were analyzed. One participant in the Positive Psychotherapy condition completed the final session but did not complete this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment
Number analyzed (Participants) | 87 | 74
units on a scale | 3.88 (0.82) | 4.07 (0.64)
Statistical Analysis 1: Comparison: Positive Psychotherapy for Smoking Cessation vs Standard Smoking Cessation Treatment; Test type: Superiority; p = 0.11, t-test, 2 sided

6. Secondary Outcome: Residual Attraction to Smoking
Description: Self-report residual attraction to smoking. Three questions are dichotomized and any positive response indicating residual attraction to smoking is coded as a 1 with any having only negative responses is coded as 0 - no residual attraction.
Time Frame: At end of treatment (4 weeks after quit date)
Population: Participants were asked these questions at the final session of counseling. Therefore only participants attending that session were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment
Number analyzed (Participants) | 88 | 74
Participants | 65 | 54
Statistical Analysis 1: Comparison: Positive Psychotherapy for Smoking Cessation vs Standard Smoking Cessation Treatment; Test type: Superiority; p = 0.90, Chi-squared

7. Secondary Outcome: Self-efficacy for Resisting Smoking
Description: Self-reported confidence in remaining abstinent from smoking. The 9-item scale uses a 1-5 response scale and the total score is the average of those 9 responses, where higher scores represent higher confidence in resisting smoking.
Time Frame: At end of treatment (4 weeks after quit date)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment
Number analyzed (Participants) | 88 | 74
units on a scale | 3.76 (1.12) | 3.80 (1.03)
Statistical Analysis 1: Comparison: Positive Psychotherapy for Smoking Cessation vs Standard Smoking Cessation Treatment; Test type: Superiority; p = 0.82, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Positive Psychotherapy for Smoking Cessation | Standard Smoking Cessation Treatment
All-Cause Mortality (participants affected / at risk) | 1/140 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/131
Other Adverse Events (participants affected / at risk) | 0/140 | 2/131
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Psychotherapy for Smoking Cessation (N=140) | Standard Smoking Cessation Treatment (N=131)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT02997657/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT02997657/SAP_001.pdf